CLINICAL TRIAL: NCT04992429
Title: Do Prostheses of SphinkeeperTM Migrate After Operation? - a Prospective Pilot Study
Brief Title: Do Prostheses of SphinkeeperTM Migrate After Operation?
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Christopher Dawoud, Principal Investigator; Dr. med. univ., Medical University of Vienna
Other Study IDs: 1814/2020
Record Dates: First submitted 2021-08-01; First posted 2021-08-05 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: SphinkeeperTM — The SphinkeeperTM includes up to 10 self-expandable prostheses, which get inserted into the intersphincteric place. They are made of inert Hyexpan (polyacrylonitrile)

SUMMARY:
32 patients who underwent sphinkeeper operation got enrolled in this study. The primary endoint is to explore the movement of the prostheses examined by manometry and ultrasound. The secondary endpoint is to find out about the functional outcome when migration of prostheses occurs and to examine differences in morphology of the sphincters after operation.

DETAILED DESCRIPTION:
The SphinkeeperTM is a new surgical procedure in order to treat refractory fecal incontinence, which includes up to ten self-expandable prostheses. These get implanted into the intersphincteric space and due to constriction of the anal canal and better contractibility continence should be improved. Because this is a new technique, there is only limited data about its clinical efficacy.

In this study, patients, aged 18-90 years, who met the inclusion criteria and have received a SphinkeeperTM operation, were enrolled. Functional outcomes and quality of life got measured by standard questionnaires before surgery and 1, 2, 3 and 6 months after surgery. Furthermore, in routine check ups patients received endoanal anorectal manometry for pressure measurement and endoanal ultrasound to determine the position of the prostheses.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 90 years, undergoing sphinkeeper operation at the Department of General Surgery, Medical University of Vienna
* Ability and willingness to understand and comply with study interventions and restrictions.
* Voluntarily signed informed consent after full explanation of the study to the participant

Exclusion Criteria:

* Any physical or mental disorder, which could interfere with the participant's safety during the clinical trial or with the study objectives
* Inability to communicate well with the investigator due to language problems or reduced mental development
* Inability or unwillingness to give written informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidates for sphinkeeper operation due to fecal incontinence will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Migration of prostheses | 6 months
  The migration got analysed by using endoanal ultrasound one, two, three and six months after surgery. The prostheses will be categorized by their position in relation to the anal canal axis.

SECONDARY OUTCOMES:
Influence of migration of the prostheses in functionality | 6 months
  Episodes of fecal incontinence and bowel habits were assessed using the Vaizey incontinence score (range 0-22, higher number means severe incontinence). It gets explored if there is a relation between migration of prostheses and worsening of incontinence.
Psychological and physical well-being | 6 months
  The psychological and physical well-being before and after operation was assessed using the SF-12 standardized questionnaire. (range 0-100; higher scores= Better quality of life)
Morphology of the anal sphincter after operation | 6 months
  Differences of the morphology before and after the operation got examined by endoanal ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Riss, Prof.MD, Study Chair — Medical University of Vienna, Head of Pelvic Floor Surgery
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
IPD can be shared just in anonymised form in case of an ethical agreement with other researchers.